CLINICAL TRIAL: NCT01892033
Title: Aerobic Exercise: Feasibility and Safety Assessment in Women Veterans With PTSD (AESAP)
Brief Title: A Pilot Exercise Study for PTSD in Women Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Geetha Shivakumar, Psychiatrist, Dallas VA Medical Center; Assistant Professor, UT Southwestern Medical Center, North Texas Veterans Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10N17
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; PTSD; Aerobic Exercise; Women; Veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aerobic Exercise (Experimental): The aerobic exercise intervention is a 12-week program consisting of four 30- to 40-minute exercise sessions of brisk walking per week.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — 12 weeks of brisk walking

SUMMARY:
The overall aim of this pilot feasibility study is to determine if 12-week moderate intensity exercise can safely alleviate posttraumatic symptoms in premenopausal women veterans.

Specific aims of the study are to;

1. Determine the feasibility, safety, and tolerability of 12-week moderate intensity exercise
2. Explore potential therapeutic benefits of 12-week moderate intensity exercise. Outcome data will include posttraumatic and depressive symptoms.
3. Explore potential therapeutic effects of a 12-week moderate intensity exercise on comorbid pain syndrome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Women veterans ages 18 and older
2. Premenopausal women of childbearing potential with a negative pregnancy test
3. DSM IV-TR confirmed PTSD related to any traumatic event as measured by Clinician Administered PTSD Scale (CAPS) with a CAPS score of at least 45
4. Relatively low sedentary life style
5. Existing psychotropic medications are allowed if on a stable dose
6. Evidence-based psychotherapy (e.g. Cognitive Processing Therapy or Prolonged Exposure) is not allowed to start of the study. However supportive or educational groups that are not PTSD-focused are allowed.

Exclusion Criteria:

1. Other psychiatric diagnoses including bipolar disorder, schizophrenia, schizoaffective disorder, active substance dependence/abuse (use in the past 1 month), obsessive-compulsive disorder, and eating disorders.Comorbid major depressive disorder, dysthymia and generalized anxiety disorders are not excluded.
2. Serious psychopathology
3. Actively suicidal or homicidal
4. Psychiatric hospitalization within the past 30 days
5. Active medical conditions that preclude the use of aerobic exercise such as uncontrolled hypertension, active musculoskeletal degenerative conditions, and symptomatic cardiovascular or respiratory conditions.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Clinician Administered Posttraumatic Stress Disorder Scale (CAPS) | Changes from baseline to week 12.

SECONDARY OUTCOMES:
PTSD Checklist | Changes from baseline to week 12.
Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) | Changes from baseline to week 12.
Pain Scale | Changes from baseline to week 12.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | Changes from baseline to week 12.
Safety (Monitoring for common side effects associated with aerobic exercise and adverse events). | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geetha Shivakumar, M.D., M.S., Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Shivakumar G, Anderson EH, Suris AM, North CS. Exercise for PTSD in Women Veterans: A Proof-of-Concept Study. Mil Med. 2017 Nov;182(11):e1809-e1814. doi: 10.7205/MILMED-D-16-00440. PMID 29087845